CLINICAL TRIAL: NCT06539533
Title: Efficacy of Pilates Training on Dynamic Balance in Flexible Flat Feet
Brief Title: Pilates on Dynamic Balance in Flexible Flat Feet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nora Mohamed Badran, professor of physical therapy basic science departement, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/005435
Record Dates: First submitted 2024-07-28; First posted 2024-08-06 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Flexible Flatfoot
MeSH Terms: conditions — Flatfoot | interventions — Exercise Movement Techniques

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental group):22 subjects (Experimental): 22 subjects will receive Pilates training. twice a week for 5 consecutive weeks, with The duration of Pilates is 30 minutes. 10 repetitions for each exercise with 10 seconds of rest between each Pilates.And short feet exercises daily 3 minutes per time, for a total of five weeks
  Interventions: Other: pilates training
- Group B (control group):22 subjects (Active Comparator): 22 subjects will receive short feet exercise daily 3 minutes per time for a total of five weeks.
  Interventions: Other: pilates training

INTERVENTIONS:
Other: pilates training — The Pilates that will be used in this study are articulating bridge, Hundreds, Plank , rolls up, one leg stretch, lift leg supine.
  Other Names: short feet exercises

SUMMARY:
Flexible flatfoot is one of the most common types of flatfeet. It has an arch that is present in open kinetic chain and lost in closed kinetic chain Balance is defined as the process that maintains the center of gravity within the body's support base.

Pilates exercises is a whole body conditioning program which was initially used for managing low back pain and improving balance in elderly. Now-a-days it is used for posture correction and fitness training.

DETAILED DESCRIPTION:
Individuals with flatfeet are more unstable when compared with normal individuals during quiet standing. About 10% to 25% of population exhibits a flat foot to varying degrees. In clinical practice, some subjects become symptomatic with feet pain or lower extremity soreness and limitation in their functional activities such as limitation of long-distance walking or running and high-impact sports.Patients with flexible flat feet have poorer static and dynamic balance than healthy individuals. Taking into consideration effect of flat feet on body alignment, the implication of flat feet on balance have received little attention to date Pilates is an individual body-based exercise, it has an advantage in that exercise load can be controlled according to the body's center of balance.Pilates based exercise works on the principles of trunk stability, also known as "core stability". "Core is described as a box, with the abdominals (transversus) in front, paraspinals (multifidus) in back, diaphragm in top and pelvic floor at the bottom". Pilates is a popular form of exercise training program which includes series of stretching and strengthening exercises with proper trunk control and breathing.

ELIGIBILITY:
Inclusion Criteria:

1. Subject's age ranged from 18-21 years old
2. Subjects had bilateral pronated feet posture according to the Navicular Drop Test by Brody method: normal feet (between five and nine mm of navicular drop), a pronated foot (more than 10 mm of navicular drop)
3. Body Mass Index (MBI) ranged from 18.5 to 25 kg/ m2

Exclusion Criteria:

* 1-Repeated lower extremity injuries as fractures or deformities. 2-History of surgery to the lower extremity. 3- Any neurological deficit affecting balance. 4-Any medication can affect the balance. 5- pregnant and breast feeding females

Ages: 18 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
dynamic balance | 6months
  is the ability to remain standing and stable while performing movements or actions that require displacing or moving oneself. In this way, each time that we take a step in any direction, we will be testing this type of balance. And, of course, the ability to walk requires its continuous use.
  Balance check 636 device (Dr Wolff, Arnsberg, Germany)for assessment of dynamic balance in each subject individually

SECONDARY OUTCOMES:
quialty of life | 6months
  sense of wellbeing embracing the physical, psychological, social, and spiritual state. • Foot function index Questionnaire (FFI) for quality of life assessment.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physical Therapy, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No